CLINICAL TRIAL: NCT02712801
Title: Antiretroviral Regime for Viral Eradication in Newborns After Intervention Failure of Mother-to-child Transmission of HIV
Brief Title: Antiretroviral Regime for Viral Eradication in Newborns
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Center for Women and Children's Health, China CDC (Other Government)
Collaborators: National Center for AIDS/STD Control and Prevention, China CDC (Other Government); Maternal and Child Health Hospital of Yunan Province (Unknown); Maternal and Child Health Hospital of Sichuan Province (Unknown); Maternal and Child Health Hospital of Guangxi Province (Unknown); Maternal and Child Health Hospital of Xinjiang Uygur Autonomous Region (Unknown); Guangdong Provincial Maternal and Child Health Hospital (Other)
Responsible Party: Principal Investigator, Xi JIN, Deputy Director, National Center for Women and Children's Health, China CDC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015ZX10001001
Record Dates: First submitted 2016-03-14; First posted 2016-03-18 (Estimated); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: HIV/AIDS and Infections
Keywords: HIV; antiretroviral treatment; child; testing
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Infections | interventions — Zidovudine; Nevirapine; Lamivudine; Lopinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): Children will receive antiretroviral treatment (ART) until 6 weeks old after birth. For the first two weeks, Zidovudine (AZT), Lamivudine (3TC) and Nevirapine (NVP) will be used. When the child is 2 weeks old, the regimen will be adjusted and Nevirapine (NVP) will be replaced by Lopinavir/ritonavir (LPV/r). Early infant diagnosis and other relevant testing will be performed to monitor children's HIV infection status. If the child is not infected, ART will be stopped when he/she reaches 6 weeks old. Otherwise, the treatment will be continued.
  Interventions: Drug: Zidovudine; Drug: Nevirapine; Drug: Lamivudine; Drug: Lopinavir/ritonavir
- Control group (Active Comparator): Children will receive routine prevention of mother-to-child transmission of HIV services. Nevirapine (NVP) or Zidovudine (AZT) will be administrated to them until 6 weeks old after birth. Early infant diagnosis services will be provided when the child is 6 weeks old and repeated when 3 months old. Children with HIV infection will be referred to receive routine HIV infection treatment.
  Interventions: Drug: Zidovudine; Drug: Nevirapine

INTERVENTIONS:
Drug: Zidovudine — Dose will be adjusted according to the child's weight.
  Other Names: AZT
Drug: Nevirapine — Dose will be adjusted according to the child's weight.
  Other Names: NVP
Drug: Lamivudine — Dose will be adjusted according to the child's weight.
  Other Names: 3TC
  Arms: Intervention group
Drug: Lopinavir/ritonavir — Dose will be adjusted according to the child's weight.
  Other Names: LPV/r
  Arms: Intervention group

SUMMARY:
This is a multi-center, randomized, controlled, open clinical trial. The trial will be carried out in five provinces in China. Pregnant women with HIV infection and at high risk of mother-to-child transmission of HIV will be identified. Their newborn babies who are at high risk HIV infection will be recruited and randomized into intervention and control groups. Children in intervention groups will receive ART and intensive HIV testing after birth. Children in control group will receive routine prevention of mother-to-child transmission services. All the included children will be followed up and their development and infection status will be recorded and compared.

ELIGIBILITY:
Inclusion Criteria:

* children whose mother with HIV infection
* children whose mother received antiretroviral drugs after 36 gestational weeks or received no drugs before delivery
* live birth

Exclusion Criteria:

* birth weight is less than 2000g
* Apgar score is less than 3 at 1 minute after birth or less than 6 at 5 minute after birth .

Ages: 0 Days to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
HIV infection in children | 0-18 months old
  Number of children diagnosed with HIV infection
Functional HIV cure in children | 0-36 months old
  Number of children with functional HIV cure

SECONDARY OUTCOMES:
Mortality | 0-36 months old
  Number of children died
ART regime for HIV exposed children at high risk of infection | 0-36 months old
  ART regime to be used for functional HIV cure in children
Testing algorithm for early infant diagnosis of HIV | 0-4 weeks old
  Testing methods and algorithm for HIV exposed infants

CONTACTS AND LOCATIONS:
Overall Officials: Xi Jin, M.D., Principal Investigator — National Center for Women and Children's Health, China CDC
Locations (5):
- China (5):
  - Maternal and Child Health Hospital of Guangdong Province, Guangzhou, Guangdong
  - Maternal and Child Health Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Maternal and Child Health Hospital of Sichuan Province, Chengdu, Sichuan
  - Maternal and Child Health Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - Maternal and Child Health Hospital of Yunan Province, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No